CLINICAL TRIAL: NCT02829970
Title: Behavioral Activation To Reduce Problem Alcohol Use In College Students With ADHD
Brief Title: Helping College Students With ADHD Lead Healthier Lifestyles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34AA022133-01A1 (NIH)
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Alcohol-Related Disorders; Substance-Related Disorders
Keywords: Attention Deficit Hyperactivity Disorder; Alcohol-Related Disorders; Substance-Related Disorders; Motivational Interviewing; Behavior Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Alcohol-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SUCCEEDS Program (Experimental): Participants will meet individually with a research team member for three weekly sessions, two bi-weekly sessions, and complete 1-month and 3-month post treatment follow-ups. Participants will be engaged about personalized alcohol feedback and identify life values and specific activities important to those values.
  Interventions: Behavioral: SUCCEEDS Program
- Living a Healthy College Lifestyle (Active Comparator): Participants will meet individually with a research team member for three weekly sessions, two bi-weekly sessions, and complete 1-month and 3-month post treatment follow-ups. Participants will engage in discussion focused on experiences as an emerging adult.
  Interventions: Behavioral: Living a Healthy College Lifestyle

INTERVENTIONS:
Behavioral: SUCCEEDS Program — Participants will receive ADHD Psychoeducation, Brief Motivational Interviewing (BMI) and Behavioral Activation for Attention & Alcohol Disorders (BAAAD).
  Arms: SUCCEEDS Program
Behavioral: Living a Healthy College Lifestyle — Participants will receive ADHD Psychoeducation, BMI and Supportive Counseling (SC).
  Arms: Living a Healthy College Lifestyle

SUMMARY:
There are currently no published randomized controlled studies examining psychosocial interventions for college students with ADHD, and none specifically targeting AUDs in this population at any age, despite the clear indication from emerging research of the need for such interventions. In the current study, the investigators will develop BA-based treatment intended to increase involvement in healthy, goal-directed activities (e.g., academic, recreational or social activities) and to reduce problematic drinking behaviors and other risk behaviors (e.g., unsafe sex) among college students with ADHD (Behavioral Activation for Attention & Alcohol Disorders; BAAAD). Finalized treatment manuals, altered based on focus group feedback, will be tested in a stage I randomized controlled trial (RCT) among 80 college students randomized to BMI + BAAAD or BMI + supportive counseling (SC). The investigators expect that BMI + BAAAD will be successful with college students with ADHD, in terms of decreasing the escalation of problematic alcohol use behaviors, as compared to BMI + SC. This treatment development study will set the stage for larger-scale RCTs.

DETAILED DESCRIPTION:
College students with Attention-Deficit/Hyperactivity Disorder (ADHD) are particularly vulnerable to problematic alcohol use (e.g., excessive alcohol consumption, failure to meet responsibilities because of drinking, or injury to self or others as a result of drinking) given their developmentally-inappropriate levels of inattention, hyperactivity and impulsivity, combined with the lifestyle associated with life on a college campus (including increased access to alcohol, decreased structure and parental supervision). Prior research demonstrates elevated rates of alcohol related problems and disorders (AUDs) among college students with ADHD; 47% of college students with ADHD meet lifetime criteria for alcohol abuse and 23% meet criteria for dependence, as compared to 12% and 6% of college students from the general population, respectively. There are currently no published randomized controlled studies examining psychosocial interventions for college students with ADHD, and none specifically targeting AUDs in this population at any age, despite the clear indication from emerging research of the need for such interventions. Moreover, brief motivation-based alcohol interventions (BMIs) that generally have been successful for college students show limited benefits among individuals with elevated impulsivity and poor self-regulation, both hallmarks of ADHD, calling for the need to modify BMIs for this vulnerable group. Thus, it is crucial to determine core treatment components that are efficacious for treating AUDs and that are developmentally-appropriate for college students with ADHD and designed in a manner which promotes transportability to the university counseling center setting. Behavioral activation (BA) is a brief behavioral approach that aims to increase individuals' contact with valued environments through systematic efforts to increase rewarding experiences, enjoyment of daily activities, and goal-directed behaviors. BA has been successfully applied to substance users in a range of settings, including college students with problematic drinking patterns. Importantly, BA has clear relevance for addressing ADHD-related executive functioning deficits, which may be associated with an increased propensity for engagement in problematic alcohol use. Further, BA teaches individuals to engage in healthy, goal-directed rewarding behaviors (e.g., academic, recreational or social activities), rather than relying on drinking to provide immediate rewards. Finally, BA is a highly adaptable intervention approach. In the current study, the investigators will develop BA-based treatment intended to increase involvement in healthy, goal-directed activities (e.g., academic, recreational or social activities) and to reduce problematic drinking behaviors and other risk behaviors (e.g., unsafe sex) among college students with ADHD (Behavioral Activation for Attention & Alcohol Disorders; BAAAD). This treatment will be developed in collaboration with the University Counseling Center, to ensure its applicability within this setting, utilizing focus group methodology with Center staff. Finalized treatment manuals, altered based on focus group feedback, will be tested in a stage I randomized controlled trial (RCT) among 80 college students randomized to BMI + BAAAD or BMI + supportive counseling (SC). The investigators expect that BMI + BAAAD will be successful with college students with ADHD, in terms of decreasing the escalation of problematic alcohol use behaviors, as compared to BMI + SC. This treatment development study will set the stage for larger-scale RCTs.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-24 years old
* Be enrolled full-time at University of Maryland - College Park (UMCP) as an undergraduate student
* Be fluent in English
* Live independently from their parents
* Meet full Diagnostic and Statistical Manual - 5th Edition (DSM-5) criteria for ADHD
* Meet cutoffs on AUDIT

Exclusion Criteria:

* Bipolar disorder or current psychosis, which would require more immediate/intensive treatment
* Current engagement in psychosocial therapy thought to interfere with this study (including participation in other treatment studies on campus)
* Suicidal risk that would place the individual at risk beyond the safety procedure available from the research team

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2015-09; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Brief Young Adult Alcohol Consequences Questionnaire 30 Day | Baseline, Post-Treatment (Week 5), 1 Month Follow-up (Week 9), 3 Month Follow-Up (Week 17)
  Changes in problematic drinking behaviors

SECONDARY OUTCOMES:
Barkley Functional Impairment Scale-Self Report | Baseline, Post-Treatment (Week 5), 1 Month Follow-up (Week 9), 3 Month Follow-Up (Week 17)
  Changes in functional impairment
Alcohol Use Disorders Identification Test | Baseline, Post-Treatment (Week 5), 1 Month Follow-up (Week 9), 3 Month Follow-Up (Week 17)
  Changes in problematic drinking behaviors
Beck Depression Inventory-II | Baseline, Week 1, Week 2, Week 3, Post-Treatment (Week 5), 1 Month Follow-up (Week 9), 3 Month Follow-Up (Week 17)
  Changes in depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Chronis-Tuscano, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: No